CLINICAL TRIAL: NCT05185297
Title: Recreational Futsal as a Coadjuvant in Male Adults With Controlled Hypertension - a Randomized Controlled Trial
Brief Title: Recreational Futsal for Controlled Hypertension
Acronym: HyperFut
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Institute of Maia (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Susana Cristina Araújo Póvoas, Associated Professor, University Institute of Maia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UMSFRH/BD/143729/2019
Record Dates: First submitted 2021-12-20; First posted 2022-01-11 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Hypertension,Essential; Hypertension; Blood Pressure Disorders; Blood Pressure
Keywords: futsal; controlled hypertension; recreational futsal; soccer; football
MeSH Terms: conditions — Essential Hypertension; Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blood analysis, maximum oxygen consumption and DEXA scans will have blinded outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): Participants will continue with standard care provided by the family physician.
- Recreational Futsal, plus standard care (Experimental): Participants will participate in 2-3 weekly one hour sessions of Recreational Futsal, during 3 months, while maintaining standard care provided by the family physician.
  Interventions: Other: Recreational Futsal

INTERVENTIONS:
Other: Recreational Futsal — Participants will participate in 2-3 weekly one hour sessions of Recreational Futsal, during 3 months, while maintaining standard care provided by the family physician.
  Arms: Recreational Futsal, plus standard care

SUMMARY:
Arterial hypertension (HT) was the leading global contributor for premature deaths in 2015. Its treatment includes medication and lifestyle changes, namely diet and regular exercise, which has shown to have an inverse relationship with arterial HT.

Recreational soccer (RS) has proven to be a non-pharmacological treatment for several chronic conditions, including arterial HT, with meaningful decreases on blood pressure (BP). Recreation futsal (RF) is expected to elicit comparable BP changes to RS considering that it imposes similar physical and physiological demands.

However, the effects of RF on BP and other cardiovascular markers have not been previously investigated in participants only with controlled arterial HT. Furthermore, acute BP changes and double product elicited by this exercise modality were never described.

Therefore, the main purpose of this study is to assess if RF is an effective coadjuvant intervention for BP control in adults with controlled arterial HT. Secondary purposes are: i) to determine the impact of RF on other cardiovascular markers; ii) to describe the acute BP changes and the double product elicited by RF; and iii) to assess the impact of 1 month of detraining on BP and other cardiovascular markers (4 months).

DETAILED DESCRIPTION:
Statistical analysis:

The efficacy of the intervention will be assessed by comparing the differences between groups at follow-up, adjusted for the outcome baseline values, systolic blood pressure, maximum oxygen consumption and age (ANCOVA).

Intention-to-treat approach will be the main analysis. The missing data will be imputed by using multiple linear regression.

A per protocol analysis will also be performed (intervention group: attendance of at least 62.5% of the training sessions; control group: participants that did not engage in regular and supervised physical exercise or had an increase in dose or number of antihypertensive medication).

The significance level will be set at 5%.

Randomization:

Stratified by baseline systolic blood pressure and maximum oxygen consumption.

Contingency plan:

If the recruitment rate is below than expected, potential measures are to include: i) 30-35- and 60-65-year-old participants; ii) participants with pre-hypertension or uncontrolled hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Medicated controlled hypertension, with habitual SBP below 140 mmHg and DBP below 90 mmHg;
* Males with 35-60 years;
* Not being engaged in regular and supervised physical exercise in the last 6 months;
* Medical clearance;
* Vaccinated against SARS-COV-2.

Exclusion Criteria:

* Cardiovascular disease (heart failure), cerebrovascular disease, advanced retinopathy or kidney failure;
* Resistant hypertension;
* History of cardiovascular event.

Ages: 35 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Between-groups differences in systolic blood pressure | 3 months
  Casual (resting) measures of systolic blood pressure (mmHg) will be measured in triplicate over the brachial artery of the non-dominant arm after 5 minutes of quiet rest, with 1 minute of recovery between each measure, using an automated oscillometric sphygmomanometer.
Between-groups differences in diastolic blood pressure | 3 months
  Casual (resting) measures of diastolic blood pressure (mmHg) will be measured in triplicate over the brachial artery of the non-dominant arm after 5 minutes of quiet rest, with 1 minute of recovery between each measure, using an automated oscillometric sphygmomanometer.

SECONDARY OUTCOMES:
Between-groups differences in systolic blood pressure | 4 months
  Casual (resting) measures of systolic blood pressure (mmHg) will be measured in triplicate over the brachial artery of the non-dominant arm after 5 minutes of quiet rest, with 1 minute of recovery between each measure, using an automated oscillometric sphygmomanometer.
Between-groups differences in diastolic blood pressure | 4 months
  Casual (resting) measures of diastolic blood pressure (mmHg) will be measured in triplicate over the brachial artery of the non-dominant arm after 5 minutes of quiet rest, with 1 minute of recovery between each measure, using an automated oscillometric sphygmomanometer.
Between-groups differences in mean blood pressure | 3 months
  Casual (resting) blood pressure (mmHg) will be measured in triplicate over the brachial artery of the non-dominant arm after 5 minutes of quiet rest, with 1 minute of recovery between each measure, using an automated oscillometric sphygmomanometer.
Between-groups differences in mean blood pressure | 4 months
  Casual (resting) blood pressure (mmHg) will be measured in triplicate over the brachial artery of the non-dominant arm after 5 minutes of quiet rest, with 1 minute of recovery between each measure, using an automated oscillometric sphygmomanometer.
Between-groups differences in total cholesterol | 3 months
  Will be analysed using standardised methods, using relevant commercial enzymatic test kits.
Between-groups differences in total cholesterol | 4 months
  Will be analysed using standardised methods, using relevant commercial enzymatic test kits.
Between-groups differences in high-density lipoprotein cholesterol | 3 months
  Will be analysed using standardised methods, using relevant commercial enzymatic test kits.
Between-groups differences in high-density lipoprotein cholesterol | 4 months
  Will be analysed using standardised methods, using relevant commercial enzymatic test kits.
Between-groups differences in low-density lipoprotein cholesterol | 3 months
  Will be analysed using standardised methods, using relevant commercial enzymatic test kits.
Between-groups differences in low-density lipoprotein cholesterol | 4 months
  Will be analysed using standardised methods, using relevant commercial enzymatic test kits.
Between-groups differences in triglycerides | 3 months
  Will be analysed using standardised methods, using relevant commercial enzymatic test kits.
Between-groups differences in triglycerides | 4 months
  Will be analysed using standardised methods, using relevant commercial enzymatic test kits.
Between-groups differences in glycosylated hemoglobin | 3 months
  Will be analysed using standardised methods, using relevant commercial enzymatic test kits.
Between-groups differences in glycosylated hemoglobin | 4 months
  Will be analysed using standardised methods, using relevant commercial enzymatic test kits.
Between-groups differences in resting heart rate | 3 months
  Number of heart beats per minute, measured by heart rate monitors.
Between-groups differences in resting heart rate | 4months
  Number of heart beats per minute, measured by heart rate monitors.
Between-groups differences in maximum oxygen consumption | 3 months
  Determined by pulmonary gas exchange measurements.
Between-groups differences in maximum oxygen consumption | 4 months
  Determined by pulmonary gas exchange measurements.
Between-groups differences in aerobic performance (Yo-Yo Intermittent Endurance Level 1 Test) | 3 months
  Number of meters covered.
Between-groups differences in aerobic performance (Yo-Yo Intermittent Endurance Level 1 Test) | 4 months
  Number of meters covered.
Between-groups differences in body mass index | 3 months
  Defined as a person's weight in kilograms divided by the square of the person's height in metres (kg/m2)
Between-groups differences in body mass index | 4 months
  Defined as a person's weight in kilograms divided by the square of the person's height in metres (kg/m2)
Between-groups differences in bone density (measured by DEXA in g/cm2) | 3 months
  bone density measured by Dual Energy X-ray Absorptiometry. Bone mineral density is expressed as absolute values (g / cm2 - grams of bone mineral content per area or analyzed bone cm2).
Between-groups differences in bone density (measured by DEXA in g/cm2) | 4 months
  bone density measured by Dual Energy X-ray Absorptiometry. Bone mineral density is expressed as absolute values (g / cm2 - grams of bone mineral content per area or analyzed bone cm2).
Between-groups differences in bone content (measured by DEXA in grams) | 3 months
  bone density measured by Dual Energy X-ray Absorptiometry. Bone mineral density is expressed as absolute values (grams)
Between-groups differences in bone content (measured by DEXA in grams) | 4 months
  bone density measured by Dual Energy X-ray Absorptiometry. Bone mineral density is expressed as absolute values (grams)
Between-groups differences in lean mass (measured by DEXA in kg) | 3 months
  measured by Dual Energy X-ray Absorptiometry (kg)
Between-groups differences in lean mass (measured by DEXA in kg) | 4 months
  measured by Dual Energy X-ray Absorptiometry (kg)
Between-groups differences in body fat (measured by DEXA in %) | 3 months
  measured by Dual Energy X-ray Absorptiometry (%)
Between-groups differences in body fat (measured by DEXA in %) | 4 months
  measured by Dual Energy X-ray Absorptiometry (%)
Between-groups differences in body mass (measured by DEXA in kg) | 3 months
  measured by Dual Energy X-ray Absorptiometry (kg)
Between-groups differences in body mass (measured by DEXA in kg) | 4 months
  measured by Dual Energy X-ray Absorptiometry (kg)
Between-groups differences in postural balance | 3 months
  measured by a modified Flamingo test
Between-groups differences in postural balance | 4 months
  measured by a modified Flamingo test
Between-groups differences in lower body strength | 3 months
  measured by a counter-movement jump test
Between-groups differences in lower body strength | 4 months
  measured by a counter-movement jump test
Between-groups differences in quality of life | 3 months
  measured by WHOQOL-BREF questionnaire
Between-groups differences in quality of life | 4 months
  measured by WHOQOL-BREF questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Susana Póvoas, PhD, Principal Investigator — University of Maia
Locations (1):
- University of Maia, Maia, Portugal

IPD SHARING:
Plan to Share IPD: No